CLINICAL TRIAL: NCT03336112
Title: Internet-delivered Cognitive Behavioral Therapy for Treatment of Cardiac Anxiety in Patients With Non-cardiac Chest Pain - a Randomized Controlled Study
Brief Title: Internet-delivered CBT for Patients With NCCP
Acronym: IKSIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Ghassan Mourad, Senior lecturer, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-CBT for NCCP
Record Dates: First submitted 2017-10-25; First posted 2017-11-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Non-cardiac Chest Pain; Cardiac Anxiety
Keywords: Non-cardiac chest pain; Psychological distress; I-CBT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 5 weeks guided internet-delivered cognitive behavioral therapy program The program consists of psychoeducation, exposure to physical activity, and awareness (mindfulness) training.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy (I-CBT)
- Control group (Active Comparator): Information program delivered by the Internet during 5 weeks.
  Interventions: Other: Information program

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioral therapy (I-CBT) — The intervention (I-CBT) will consist of 5 weeks of Internet-delivered cognitive behavioral therapy using three main parts. The first is psychoeducation that aims to educate the patients about chest pain and other causes than the cardiac ones. The other part concerns avoidance and exposure. This includes exposing the patients to physical activities that patients perceive as a threat to the heart. The third part contains awareness (mindfulness) training to teach the patients to have contact with the present moment despite chest pain and not trying to avoid it.
  Arms: Intervention group
Other: Information program — Information program delivered by the Internet during 5 weeks.
  Arms: Control group

SUMMARY:
Non-cardiac chest pain (NCCP) is common and has substantial impact on patients' psychological wellbeing, quality of life and healthcare use. Although cardiac diagnosis is 'ruled out', many patients think they have an undetected cardiac disease (i.e. they suffer cardiac anxiety) as no other explanation is offered. They therefore avoid activities that they believe might be harmful to their heart, leading to greater ill-health, and increased healthcare use and societal costs. Targeting cardiac anxiety with psychological interventions might break this vicious circle and improve patient outcomes. Patients need to evaluate the way they perceive and handle their chest pain, which can be done with cognitive behavioral therapy (CBT).

The aim of this study is therefore to evaluate the short- and long-term effects of an Internet-delivered CBT (I-CBT) program on psychological distress and other patient-reported outcomes in patients with NCCP. A second aim is to explore factors related to implementation of I-CBT in clinical care. The study has a randomized controlled design comparing I-CBT with Internet-delivered information program. Quantitative methods will be used to evaluate the effectiveness of the I-CBT program. Implementation issues will be evaluated from the perspectives of patients, healthcare professionals and policymakers using qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 healthcare visits due to NCCP during the last 6 months
* patients suffering from cardiac anxiety (score ≥ 24 on the Cardiac Anxiety Questionnaire-CAQ)

Exclusion Criteria:

* language difficulties
* not able to perform physical activity/exercise due to physical constraints
* patients with severe depressive symptoms
* patients with acute ischemic heart disease
* patients with no access to computer/tablet and/or Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiac anxiety | 12 months after end of intervention
  Cardiac Anxiety Questionnaire (CAQ) will be used before and after the intervention (5 weeks), and 3, 6, 12 months after the end of the intervention to assess changes related to intervention. The CAQ consists of 18 items and a score range between 0 and 72. The higher scores the greater cardiac anxiety.

SECONDARY OUTCOMES:
Fear of body sensations | 12 months after end of intervention
  Body Sensations Questionnaire will be used before and after the intervention (5 weeks), and 3, 6, 12 months after the end of the intervention to assess changes related to intervention. The questionnaire comprises 17 items with scores ranging between 17 and 85 and the higher scores the greater fear of body sensations.
Depressive symptoms | 12 months after end of intervention
  Patient Health Questionnaire-9 will be used before and after the intervention (5 weeks), and 3, 6, 12 months after the end of the intervention to assess changes related to intervention. This questionnaire comprises 9 items with scores ranging between 0 and 27. Higher scores indicate higher levels of depressive symptoms. A cut-off of 10 demonstrates moderate levels and will be used in this study.
Health-related quality of life | 12 months after end of intervention
  EuroQol-5D (EQ-5D) will be used before and after the intervention (5 weeks), and 3, 6, 12 months after the end of the intervention to assess changes related to intervention. The EQ-5D includes five dimensions of Health-related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels corresponding to: no problems, slight problems, moderate problems, severe problems and extreme problems/unable. The questionnaire also includes an EQ-VAS, which is a visual analogue scale ranging from 0 (worst health you can imagine) to 100 (best health you can imagine).
Chest pain frequency | 12 months after end of intervention
  Self-developed open questions will be used before and after the intervention (5 weeks), and 3, 6, 12 months after the end of the intervention to assess changes in chest pain related to intervention.
Healthcare use | 12 months after end of intervention
  Care Data Warehouse (Register), data will be collected 12 months after the end of the intervention to assess changes related to intervention.
Societal costs | 12 months after end of intervention
  Cost per patient register and Social Insurance Office register, data will be collected 12 months after the end of the intervention to assess changes related to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Mourad, PhD, Study Chair — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eriksson-Liebon M, Westas M, Johansson P, Mourad G. Long-term effects and predictors of change of internet-delivered cognitive behavioural therapy on cardiac anxiety in patients with non-cardiac chest pain: a randomized controlled trial. BMC Psychiatry. 2024 Mar 19;24(1):216. doi: 10.1186/s12888-024-05661-y. PMID 38504157
- [Derived] Eriksson-Liebon M, Lundgren J, Rytterstrom P, Johansson P, Mourad G. Experience of internet-delivered cognitive behavioural therapy among patients with non-cardiac chest pain. J Clin Nurs. 2023 Jul;32(13-14):4060-4069. doi: 10.1111/jocn.16565. Epub 2022 Oct 27. PMID 36303332
- [Derived] Mourad G, Eriksson-Liebon M, Karlstrom P, Johansson P. The Effect of Internet-Delivered Cognitive Behavioral Therapy Versus Psychoeducation Only on Psychological Distress in Patients With Noncardiac Chest Pain: Randomized Controlled Trial. J Med Internet Res. 2022 Jan 28;24(1):e31674. doi: 10.2196/31674. PMID 35089153